CLINICAL TRIAL: NCT06168734
Title: A Phase 3 Study to Evaluate Cefepime-taniborbactam Compared to Meropenem in Adults With Ventilator Associated Bacterial Pneumonia (VABP) or Ventilated Hospital Acquired Bacterial Pneumonia (vHABP)
Brief Title: Cefepime-taniborbactam vs Meropenem in Adults With VABP or Ventilated HABP
Acronym: CERTAIN-2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study suspended
Sponsor: Venatorx Pharmaceuticals, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VNRX-5133-301; 2022-502682-16 (EudraCT Number)
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Ventilator-associated Pneumonia; Hospital-acquired Pneumonia
Keywords: Ventilated Pneumonia; Hospital Acquired Pneumonia; Bacterial Pneumonia; VABP; vHABP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Pneumonia, Bacterial | interventions — Meropenem

STUDY DESIGN:
Intervention Model Description: The study will randomize approximately 316 patients with vHABP or VABP into 2 groups in a 1:1 ratio (158 patients to cefepime-taniborbactam; 158 patients to meropenem).
Who Masked: Participant, Investigator
Masking Description: A double-blind design is used to maintain blinding for all personnel involved with the evaluation of patient efficacy and safety during the study. With the exception of the unblinded pharmacist or designee, unblinded study monitors and scientists conducting plasma assays and analyses for PK assessments, the sponsor, investigator, patient, and study site staff, will remain blinded to study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cefepime-taniborbactam (Experimental): cefepime-taniborbactam (2g/0.5g) IV every 8 hours.
  Interventions: Drug: Cefepime-taniborbactam
- Meropenem (Active Comparator): Comparator: meropenem (2g) IV every 8 hours.
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Cefepime-taniborbactam — Cefepime-taniborbactam administered 2.5g q8h intravenously (IV) over a 4-hour period for 7 days to 14 days at the investigator's discretion. Dose adjustments for renal function may apply.
  Arms: Cefepime-taniborbactam
Drug: Meropenem — Meropenem will be administered 2g q8h IV over 4 hours for 7 days to 14 days at the investigator's discretion. Dose adjustments for renal function may apply.
  Arms: Meropenem

SUMMARY:
This is a Phase 3, randomized, multicenter, double-blind, non-inferiority study to evaluate the efficacy and safety of cefepime-taniborbactam compared to meropenem in patients ≥ 18 years of age with ventilated HABP or VABP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 years of age.
* The patient or patient's legally authorized/acceptable representative (LAR) has voluntarily signed and dated the IRB/IEC approved ICF
* Meets the clinical diagnosis of ventilated HABP or VABP
* Have at least one of the following clinical criteria:

  1. New onset or worsening of pulmonary symptoms and signs
  2. New onset or worsening of purulent respiratory secretions
  3. Hypoxemia
  4. Need for acute changes in ventilator support
* Have at least one of the following clinical criteria:

  1. Documented fever (defined as body temperature ≥ 38°C [100.4°F]
  2. Hypothermia (defined as body temperature ≤ 35°C [95°F])
  3. White blood cell (WBC) ≥10,000 cells/mm3 or ≤4,500 cells/mm3
  4. >15% immature neutrophils (bands).
* Have new or worsening infiltrate on a pulmonary imaging study that is consistent with bacterial pneumonia within 48 hours prior to randomization.
* Have a lower respiratory tract specimen sent for Gram stain and quantitative culture within 36 hours prior to the first dose of study drug.

Exclusion Criteria:

* Receipt of effective antibacterial treatment for pneumonia for a continuous duration of >24 hours during the previous 72 hours prior to randomization.
* Pneumonia known or suspected to be caused by:

  1. A bacterial pathogen resistant to meropenem, as assessed by susceptibility testing or against which either one or both study drugs lack activity
  2. Viruses, atypical bacteria, or fungi
* Use of non-study systemic gram-negative therapy.
* Confounding respiratory conditions.
* Receiving extracorporeal membrane oxygenation (ECMO).
* Patients with refractory septic shock.
* Active immunosuppression.
* Has a history of serious hypersensitivity (e.g., anaphylaxis), serious allergy, or any serious reaction to cephalosporin, penicillin, carbapenem, or other β-lactam antibiotics.
* Female patients who are pregnant.
* Patients with eGFR <10 mL/min/1.73 m2 or are receiving or starting renal replacement therapy or expected to require renal replacement therapy during the treatment phase of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ACM through Study Day 14 | Evaluated on Day 15
  The primary endpoint is ACM, a binary variable, through Study Day 14. The primary endpoint is evaluated in the ITT population and is based on the patient's survival status through Study Day 14.

SECONDARY OUTCOMES:
ACM through Study Day 28 | Evaluated on Day 29-33
  ACM through Study Day 28; analyzed in ITT and MITT analysis populations.
Safety Outcomes | From first dose up to Day 33
  Safety assessments include the incidence of TEAEs and SAEs, and discontinuation of study drug due to TEAEs.

IPD SHARING:
Plan to Share IPD: No